CLINICAL TRIAL: NCT04987567
Title: Effect of Antioxidant Docosahexaenoic Acid (DHA) Supplementation in Cystic Fibrosis Patients: A Randomized Placebo-controlled Trial
Brief Title: Effect of Antioxidant Docosahexaenoic Acid (DHA) in Cystic Fibrosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Roser Ayats-Vidal, Principal Investigator, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PED-DHA-FQ
Record Dates: First submitted 2021-06-23; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-06

CONDITIONS: Cystic Fibrosis in Children
Keywords: cystic fibrosis; Docosahexaenoic Acid; fatty acids
MeSH Terms: conditions — Cystic Fibrosis | interventions — Olive Oil

STUDY DESIGN:
Intervention Model Description: Is not a drug, is a food supplement.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antioxidant docosahexaenoic acid (DHA) (Active Comparator): Antioxidant docosahexaenoic acid (Tridocosahexaenoin-AOX ® 70%) 50mg/kg/day:
  50mg/kg/day so:
  * > = 13-17kg: 2 pearls (700mg DHA) every day, once or twice daily (od or bd)
  * > = 18-24kg: 3 pearls (1050mg DHA) every day, od or bd
  * > = 25-30kg: 4 pearls (1400mg DHA) every day, bd (2-0-2)
  * > = 31-36kg: 5 pearls (1750mg DHA) every day, bd (2-0-3)
  * > = 37-43kg: 6 pearls (2100mg DHA) every day, bd (3-0-3)
  * > = 44-49kg: 7 pearls (2450mg DHA) every day, three times a day (td) (3-1-3)
  * > = 50kg: 8 prearls (2800mg DHA) every day, td (3-2-3).
  Interventions: Dietary Supplement: ANTIOXIDANT DHA TRIGLYCERIDE (TRIDOCOSAHEXAENOINE-AOX®)
- Placebo (Placebo Comparator): Olive oil 50mg/kg/day so:
  * > = 13-17kg: 2 pearls every day, once or twice daily (od or bd)
  * > = 18-24kg: 3 pearls every day, od or bd
  * > = 25-30kg: 4 pearls every day, bd (2-0-2)
  * > = 31-36kg: 5 pearls every day, bd (2-0-3)
  * > = 37-43kg: 6 pearls every day, bd (3-0-3)
  * > = 44-49kg: 7 pearls every day, three times a day (td) (3-1-3)
  * > = 50kg: 8 prearls every day, td (3-2-3).
  Interventions: Dietary Supplement: PLACEBO (OLIVE OIL)

INTERVENTIONS:
Dietary Supplement: ANTIOXIDANT DHA TRIGLYCERIDE (TRIDOCOSAHEXAENOINE-AOX®) — Pearls of DHA (BrudyNen)
  Arms: Antioxidant docosahexaenoic acid (DHA)
Dietary Supplement: PLACEBO (OLIVE OIL) — Pearls manufactured to mimic DHA (BrudyNen).
  Arms: Placebo

SUMMARY:
This study evaluates the effect of antioxidant docosahexaenoic acid (DHA) in patients with cystic fibrosis. Half of participants will receive DHA, while the other half will receive placebo.

DETAILED DESCRIPTION:
Several studies show that patients with cystic fibrosis (CF) usually have, compared to the normal population, low levels of linoleic acid (LA) and docosahexaenoic acid (DHA) and increase in arachidonic acid (AA), which is pro-inflammatory. Normalization or modification of this fatty acid pattern (AP) could reduce chronic inflammation. The aim of this study is to assess the effect of oral supplementation with DHA for one year in pediatric patients (6-18 years) with CF, on inflammatory parameters, AP profile, lung function (spirometry) and number of exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders with a diagnosis of cystic fibrosis.
* FEV1 > 40%.
* Age between 6 and 18 years.
* Patients who grant their informed consent or whose representative grants informed consent to participate in the study.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Basal oxygen saturation <92% or household supplemental oxygen needs.
* Massive hemoptysis
* Patients who are not able to follow or who cannot be assessed in the study according to the protocol.
* Any circumstance that, at the discretion of the doctor, may involve a clinical risk or harm, the patient's participation in the study or that interferes with the evaluation of the same.
* Use of systemic glucocorticoids or in the 4 weeks prior to inclusion in the study.
* Use of non-steroidal anti-inflammatory drugs in the 2 weeks prior to inclusion in the study.
* Use of investigational drugs or participation in another clinical trial within 30 days prior to inclusion in the study or within the 5 elimination half-lives of the investigational drug.
* Be already supplementing with Omega -3, fish oil or DHA

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Fatty Acid (FA) profile (percentage) of the erythrocyte membrane at 6 and 12 months | baseline, 6 month and 12 month of treatment (end of study)
  After blood sampling, erythrocytes are separated from the plasma by centrifugation (2500 rpm for 15 min) and stored at -80ºC until analysed. The fatty acids composition are analyzed by gas chromatography.
  Fatty acid composition (SFA (saturated FA), MUFA (monoinsatured FA), PUFAs N-6 (polyunsaturated FA omega-6) and PUFAS N-3) are mesured as percentage of total fats.

SECONDARY OUTCOMES:
Change from Baseline Serum interleukins at 12 months | baseline and 12 month of treatment (end of study)
  Serum are obtained by centrifugation of blood samples and frozen at -80ºC until testing.
  Interleukins (IL)-1 β, IL-6, IL-8 and tumor necrosis factor (TNF)-α (pg/ml) are analized in serum by enzyme-linked immunosorbent assay (ELISA kits).
Change from baseline pulmonary function at 3,6 ,9 and 12 months | baseline, 3 months, 6 month, 9 months and 12 month of treatment (end of study)
  Forced expiratory volume in 1 second (FEV1) , forced vital capacity (FVC) and 25-75% of the forced vital capacity (FEF25-75%) were mesured using spirometry, calibrated daily according to standardized techniques.
  The results are expressed as the mean value of the percentage of predicted values according to height and sex and litres (L)
Number of Pulmonary exacerbation during the study year compared with previous years | 12 months prior study, 12 months of the study
  The investigators will report the number of pulmonary exacerbations during the previous year and the year of the study. To calculate the number of exacerbations, the medical records of the patients will be reviewed.
Change from baseline fecal calprotectin at the 12 months | Baseline and 12 months
  Calprotectin was measured in fecal samples of the participants.
Adverse reactions during the study | baseline, 3, 6 , 9 and 12 month of treatment (end of study)
  Frequency of occurrence of adverse events related to the study treatment: diarrhea, steatorrhea, abdominal pain, nausea, vomiting, gastroesophageal reflux, fishy taste or hemorrhage.
Change from Baseline Esputum interleukins at 6 and 12 months | baseline and 12 months
  Supernatant induced sputum were frozen at -80ºC until testing. Induced sputum Interleukins (IL)-1 β, IL-6, IL-8 and tumor necrosis factor (TNF)-α (pg/ml) were analized by enzyme-linked immunosorbent assay (ELISA kits).
Change from baseline differencial cell counts in sputum at 6 and 12 months. | baseline, 6 months and 12 monts
  An equal volume of sterile dithiothreitol (DTT), freshly diluted to 10% by the addition of sterile saline, was added to the sputum. This step was performed under a Bio-safety hood using sterile technique. The samples were then incubated in a shaking water bath at 37° C for 5-10 min, and gently mixed using a transfer pipette at 5-min intervals. The weight of the remaining sputum mixture was measured, and a further three times the volume of both DTT and phosphate-buffered saline (Dulbecco's; Gibco BRL, Grand Island, NY) were added. The mixture was incubated once again in the 37° C shaking water bath for another 5-10 min to ensure complete homogenization. Ten microliters of the homogenized sputum samples, mixed with Trypan Blue stain, was used to calculate total cell counts, using a standard hemacytometer. A further 0.25-0.50 ml of both samples was used to prepare cytospin slides for differential cell counts.
Change from baseline weight at 3, 6, 9 and 12 months | Baseline, 3,6,9 and 12 months
  Weight in kilograms (kg) were measured every 3 months. Subjects dressed only in light underwear and shoeless.
Change from baseline height at 3, 6, 9 and 12 months | Baseline, 3,6,9 and 12 months
  Height was measured with a standardised statdiometer every 3months
Change from baseline body mass index (BMI) at 3, 6, 9 and 12 months | Baseline, 3,6,9 and 12 months
  BMI was calculate every 3 months.
Change from Baseline FA ratios of the erythrocyte membrane at 6 and 12 months | baseline, 6 months and 12 months
  The next fatty acids (FA) ratios were calculated:
  Arachidonic acid /eicosapentaenoic acid (ARA/EPA) Arachidonic acid/ docosahexaenoic acid (ARA/DHA) N-3 PUFAS/ALA ( α-linolenic acid) N-6 PUFAS/LA (linoleic acid)

CONTACTS AND LOCATIONS:
Overall Officials: Roser Ayats Vidal, MD, Principal Investigator — Parc Tauli Hospital from Sabadell (Barcelona). Spain.
Locations (1):
- Parc Tauli Hospital, Sabadell, Barcelona, Spain